CLINICAL TRIAL: NCT05655689
Title: Evaluation of Antibiogram Results and Clinical Response to Prescribed Antimicrobials in Microbial Keratitis Patients
Brief Title: The Antibiogram and Outcomes of Antimicrobial Regimens in Microbial Keratitis: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Other Study IDs: ID 0106991
Record Dates: First submitted 2022-11-22; First posted 2022-12-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2022-11

CONDITIONS: Bacterial Keratitis; Fungal Keratitis; Mixed Bacterial and Fungal Keratitis; Microbial Keratitis
Keywords: Microbial keratitis; Infectious corneal ulcer; Bacterial keratitis; Fungal keratitis; Mycotic keratitis; Antibiogram; Antimicrobial resistance; Culture; Sensitivity; Fortified antibiotics eye drops; Moxifloxacin; Natamycin; Voriconazole; Prevalence; Antifungal eye drops; Bacteria; Fungi; Vancomycin; Ceftazidime; Gentamicin; Mixed bacterial and fungal keratitis
MeSH Terms: conditions — Hypersensitivity | interventions — Ophthalmic Solutions; Moxifloxacin; Ceftazidime; Gentamicins; Natamycin; Voriconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Bacterial keratitis: Microbial keratitis patients diagnosed with bacterial keratitis and treated with the empiric topical antibiotics eye drops at the usual doses for the management of bacterial keratitis, as part of routine medical care.
  Interventions: Drug: Moxifloxacin Ophthalmic 0.5% Ophthalmic Solution; Drug: Ceftazidime 5% + vancomycin 5%; Drug: Gentamicin 1.4% + vancomycin 5%
- Fungal keratitis: Microbial keratitis patients diagnosed with fungal keratitis and treated with the empiric topical antifungals eye drops at the usual doses for the management of fungal keratitis, as part of routine medical care.
  Interventions: Drug: Natamycin 5% Oph Susp; Drug: Voriconazole 1%; Drug: Natamycin 5% + voriconazole 1%
- Mixed bacterial and fungal keratitis: Microbial keratitis patients diagnosed with mixed bacterial and fungal keratitis and treated with the empiric topical antibiotics and antifungals eye drops at the usual doses for the management of mixed bacterial and fungal keratitis, as part of routine medical care.
  Interventions: Drug: Natamycin 5%+ ceftazidime 5% + vancomycin 5%; Drug: Voriconazole 1% + ceftazidime 5% + vancomycin 5%

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic 0.5% Ophthalmic Solution — In the observational study, patients treated with topical antibiotic moxifloxacin 0.5% eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: Vigamox®
  Groups: Bacterial keratitis
Drug: Ceftazidime 5% + vancomycin 5% — In the observational study, patients treated with topical fortified antibiotics ceftazidime 5% and vancomycin 5% eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: (CAZ-VAN)
  Groups: Bacterial keratitis
Drug: Gentamicin 1.4% + vancomycin 5% — In the observational study, patients treated with the topical fortified antibiotics gentamicin 1.4% and vancomycin 5% eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: (GEN-VAN)
  Groups: Bacterial keratitis
Drug: Natamycin 5% Oph Susp — In the observational study, patients treated with the topical natamycin 5% antifungal eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Groups: Fungal keratitis
Drug: Voriconazole 1% — In the observational study, patients treated with voriconazole 1% antifungal eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: Vfend®
  Groups: Fungal keratitis
Drug: Natamycin 5% + voriconazole 1% — In the observational study, patients treated with the topical natamycin 5% and voriconazole 1% antifungals eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: (NT-VRC)
  Groups: Fungal keratitis
Drug: Natamycin 5%+ ceftazidime 5% + vancomycin 5% — In the observational study, patients treated with the topical natamycin 5% and antifungal and the fortified antibiotic ceftazidime 5% and vancomycin 5% eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: (NT-CAZ-VAN)
  Groups: Mixed bacterial and fungal keratitis
Drug: Voriconazole 1% + ceftazidime 5% + vancomycin 5% — In the observational study, patients treated with the topical voriconazole 1% antifungal and the fortified antibiotics ceftazidime 5% and vancomycin 5% eye drops as part of routine medical care are observed. The investigator does not assign any specific intervention to the study participants.
  Other Names: (VRC-CAZ-VAN)
  Groups: Mixed bacterial and fungal keratitis

SUMMARY:
This study is an observational prospective cohort study which aims to generate an antibiogram and to assess the clinical responses and outcomes of microbial keratitis patients, treated with empiric topical antimicrobial therapies, with the main objective being to recommend the most effective empiric therapy. Microbial keratitis patients are attending the Cornea Outpatient Clinic at Alexandria Main University Hospital, Alexandria, Egypt.

DETAILED DESCRIPTION:
The main objective of this observational study is to recommend the most effective empiric topical antimicrobial therapy in microbial keratitis, according to the current local antimicrobial resistance data and the clinical outcomes of patients with bacterial, fungal, and mixed bacterial and fungal keratitis being treated with different empiric topical antibiotics and antifungal therapies.

In the study, test results of routinely performed culture and sensitivity on corneal scraping samples and on contact lenses in indicated severe, centrally located, and large ulcers are collected and analyzed. The sensitivity data is utilized to generate an antibiogram to describe the local prevalence of bacteria and fungi causing microbial keratitis and to investigate the prevalence of antimicrobial resistance.

Results of the culture and sensitivity are often delayed, hence empiric broad- spectrum antimicrobial therapy is ideally started after corneal scraping, until laboratory test results are obtained. Broad-spectrum empiric therapy will be modified into a more selective culture- guided therapy if the causative agent and its antimicrobial sensitivity are identified.

Empiric therapy continues in cases where the culture results are negative together with clinical improvement. Also, when patients have already been on empiric treatment before presenting to the clinic, corneal scraping and culture are not performed.

In the study, microbial keratitis patients diagnosed as either bacterial, fungal, or mixed bacterial and fungal keratitis, taking the empiric topical antimicrobials, are observed. The study investigator 's role is to observe and study the clinical responses and treatment outcomes of microbial keratitis patients who are on different empiric antimicrobial therapies as part of the routine medical care. There is no assignment of any intervention to the study participants. The investigator does not intervene, and does not prescribe, recommend, or assign any intervention to the study participants.

The clinical response of microbial keratitis patients, who are on different empiric antibiotics and antifungal eye drops, is studied by determining the primary and secondary outcomes. Measured outcomes include corneal ulcer healing, time to epithelialization, improvement in visual acuity, rates of surgical interventions and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with bacterial keratitis either clinically or by culture.
* Patients diagnosed with fungal keratitis either clinically or by culture.
* Patients diagnosed with mixed bacterial and fungal keratitis either clinically or by culture.

Exclusion Criteria:

* Patients diagnosed with corneal abrasions and non-infectious corneal ulcers.
* Patients diagnosed with acanthamoeba keratitis as a single causative agent.
* Patients diagnosed with viral keratitis as a single causative agent.
* Patients who are noncompliant to treatment.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Bacterial keratitis, fungal keratitis, and mixed bacterial and fungal keratitis patients attending the Cornea Outpatient Clinic at Alexandria Main University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Corneal ulcer healing | 4 months from participation
  An ulcer is recognized as healed when there is a lack of epithelial defect, and no infiltrates. This is detected by the routine examination under the cobalt-blue light of the slit lamp biomicroscope. The absence of fluorescein staining when fluorescein is applied to the ulcer indicates an intact epithelium.
The time to epithelialization | 4 months from participation
  The time required to re-epithelialization of the corneal ulcer is measured in days.
The antibiogram generation | 4 months from participation
  The corneal scraping culture and sensitivity test results are collected to produce the local antibiogram. Antimicrobial susceptibility is determined using the standard agar disc-diffusion method (Kirby-Bauer) by measuring the zone of inhibition. For each isolate, percentage susceptibility to the antimicrobial is calculated by dividing the number of susceptible isolates by the total number of tested isolates.

SECONDARY OUTCOMES:
The best spectacle-corrected visual acuity | 4 months from participation
  The best spectacle-corrected visual acuity (BCVA) is routinely measured using the Snellen chart. The baseline (BCVA) and the post-treatment (BCVA) are recorded as decimal values of Snellen fractions. For patients with very low vision, the semiquantitative scale of counting fingers (CF), hand motion (HM), perception of light (PL) and no perception of light (NPL) is quantified by their conversion into the equivalent decimal values using the Freiburg Visual Acuity Test (FrACT). The improvement in (BCVA) is measured by finding the difference between the post-treatment BCVA and the baseline BCVA.
Surgical interventions | 4 months from participation
  The percentage of surgical interventions is calculated. An example of surgical intervention is therapeutic penetrating keratoplasty (TKP)
Corneal perforations | 4 months from participation
  The percentage of corneal perforations is calculated. Corneal perforations are routinely tested by the Seidel test on slit lamp biomicroscope examination with cobalt blue light.
Corneal melting | 4 months from participation
  The percentage of corneal melting is calculated. Corneal melting is clinically diagnosed by the slit lamp biomicroscope examination.
Corneal opacities | 4 months from participation
  The percentage of corneal opacities is calculated. The presence of corneal opacity is detected by the slit lamp biomicroscope examination.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly M Mohamed, PhD, Principal Investigator — Associate Professor of Microbiology and Immunology, Alexandria University; Tamer H Massoud, PhD, Principal Investigator — Associate Professor of Ophthalmology, Alexandria University; Noha A Hamdy, PhD, Principal Investigator — Assistant Professor of Clinical Pharmacy, Alexandria University; Amira A Nayel, PharmD, Principal Investigator — Master's student at the Department of Clinical Pharmacy and Pharmacy Practice, Alexandria University
Locations (1):
- Cornea Outpatient Clinic at Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nayel AA, Hamdy NA, Massoud TH, Mohamed NM. A comparison of antimicrobial regimen outcomes and antibiogram development in microbial keratitis: a prospective cohort study in Alexandria, Egypt. Graefes Arch Clin Exp Ophthalmol. 2024 Jun;262(6):1865-1882. doi: 10.1007/s00417-023-06362-0. Epub 2024 Jan 19. PMID 38240778